CLINICAL TRIAL: NCT06753994
Title: Continuous Ketone Monitoring in Participants With Type 1 Diabetes (T1D) Using SGLT2 Inhibitors as Adjunctive Therapy
Brief Title: Continuous Ketone Monitoring in People With Type 1 Diabetes Using SGLT2 Inhibitors
Acronym: EmpaCKM
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Endocrinologist, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-0807
Record Dates: First submitted 2024-12-13; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; Type1diabetes; T1D
Keywords: CKM; Continous Ketone Monitoring; Empagliflozin; SGLT2i; SGLT2 inhibitors; Sodium-glucose cotransporter-2 inhibitors; Low-carb; Exercise
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity | interventions — Sodium-Glucose Transporter 2 Inhibitors; empagliflozin

STUDY DESIGN:
Intervention Model Description: This is an open- label, single-arm, outpatient study where 24 participants with type 1 diabetes will use continuous ketone monitoring for a 4-week run-in, followed by empagliflozin 2.5 mg for four weeks and then empagliflozin 10 mg for nine weeks. Participants will perform an exercise sub-study during the fourth week of the continuous ketone monitoring run-in and during the eighth week of empagliflozin 10 mg use. Certain participants will be invited to undergo a low-carbohydrate diet during the last week of empagliflozin 10 mg use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SGLT2 inhibitor dose scalation to maximum tolerated dose with Continuous Ketone Monitor (Experimental): This is a single arm study where 24 participants with T1D will use a CKM for a 4-week run-in followed by empagliflozin 2.5 mg for four weeks then empagliflozin 10 mg for nine weeks. Participants will perform an exercise sub-study during the fourth week of the CKM run-in and during the eighth week of empagliflozin 10 mg use. Certain participants will be invited to undergo a low-carb diet during the last week of empagliflozin 10 mg use.
  Interventions: Drug: SGLT-2 inhibitor

INTERVENTIONS:
Drug: SGLT-2 inhibitor — Empagliflozin is an SGLT2i that aids in blood glucose reduction through the urination of excess glucose in the context of hyperglycemia. In this study, participants will start with a dose of 2.5 mg of empagliflozin for four weeks, which will then be increased to 10 mg for the following nine weeks.
  Other Names: Empagliflozin; Sodium-glucose cotransporter-2 (SGLT2) inhibitors

SUMMARY:
Type 1 diabetes is an autoimmune disease where the body attacks the insulin-producing cells in the pancreas. In the absence of insulin, the body is unable to effectively use glucose for energy, resulting in high blood sugar levels. This leads to a lifelong need for intensive insulin therapy to manage blood sugar and prevent complications arising from elevated blood glucose levels. When insulin is low, the body produces ketone bodies. If ketone levels rise too high, they can lead to the dangerous condition known as diabetic ketoacidosis. Diabetic ketoacidosis remains a leading cause of mortality in children and young adults with type 1 diabetes.

Sodium/glucose cotransporter 2 inhibitors, such as empagliflozin, are effective in lowering blood sugar but can also increase ketone levels, raising the risk of diabetic ketoacidosis. Empagliflozin is approved for type 2 diabetes and has demonstrated benefits in type 1 diabetes, including improved blood sugar control at lower doses and reduced risks of chronic kidney disease and mortality at higher doses. However, its use in type 1 diabetes is still off-label due to the heightened risk of diabetic ketoacidosis. Using empagliflozin at a commercial dose safely is desirable to maximize its potential renal benefits in type 1 diabetes. While there are measures to monitor ketone levels, current methods, such as finger prick tests, often detect issues too late to prevent diabetic ketoacidosis. Continuous ketone monitoring offers real-time tracking of ketone levels, which could enable timely interventions to maintain safe levels. Moreover, there is currently no data on continuous ketone metrics in individuals with type 1 diabetes using sodium/glucose cotransporter 2 inhibitors.

We aim to understand the dynamics of ketone levels in people with type 1 diabetes using empagliflozin, including in challenging situations such as during exercise and low-carbohydrate diets while on sodium/glucose cotransporter 2 inhibitors. To this end, we will conduct an open- label, single-arm, outpatient study where 24 participants with type 1 diabetes will use continuous ketone monitoring for a 4-week run-in, followed by empagliflozin 2.5 mg for four weeks and then empagliflozin 10 mg for nine weeks. Participants will perform an exercise sub-study during the fourth week of the continuous ketone monitoring run-in and during the eighth week of empagliflozin 10 mg use. Certain participants will be invited to undergo a low-carbohydrate diet during the last week of empagliflozin 10 mg use. The results, if positive, may lead to i) novel long-term (6 months) data on ketone levels in those with type 1 diabetes using empagliflozin, including individuals on multiple daily injections and closed-loop therapy across a wide range of body mass index, ii) data on the relationship between empagliflozin, exercise, low-carbohydrate diets, and type 1 diabetes, and iii) the creation of important metrics for ketone thresholds that have not yet been characterized. Furthermore, we hope this preliminary study will inform future research to investigate the use of continuous ketone monitoring to allow for the safe use of higher doses of sodium/glucose cotransporter 2 inhibitors in people with type 1 diabetes.

ELIGIBILITY:
Adults ≥ 18 years old.

* A T1D diagnosis for at least one year, as per their treating physician in agreement with the investigator's judgment (confirmatory C-peptide and antibodies will not be required).
* HbA1c level of < 11% within the last six months.
* Current use of intensive insulin therapy, either multi-daily injection or closed-loop insulin pump therapy, with no plan to change during the study.
* Current use of CGM, either real-time or intermittent.
* Active avoidance of pregnancy during the trial, which includes effective contraception for any individuals of childbearing potential, who are sexually active.
* Ability to consume an average of more than 50 g of carbohydrates per day.
* Use of a compatible phone to allow for download of the CKM sensor application.

Exclusion Criteria:

* DKA or severe hypoglycemia within the last six months.
* Current or recent use of any anti-hyperglycemic agent other than insulin (≤ one month for GLP1-RA, ≤ one week for all others).
* Current or ≤ one-month use of supraphysiological doses of glucocorticoids.
* Body mass index < 20 kg/m2.
* Glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2 as per CKD-EPI formula with creatinine levels measured within the last two months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of events ≥ 0.6 mmol/L, ≥ 0.8 mmol/L ≥ 1.5 mmol/L, ≥ 3.0 mmol/L that last for more than one hour | 17 weeks
  Number of events at each range that last for more than one hour. This will be compared between i) each study period (run-in, 2.5 mg, 10 mg etc) and ii) the first week and the remaining weeks for each study period

OTHER OUTCOMES:
Beta-hydroxybutyrate level (mmol/L) | 17 weeks
  Mean, median, standard deviation and Coefficient of variation (mean/standard deviation): 24-hour, daytime (6h00-24h00), and night-time (24h00-6h00). This will be compared between each study period (run-in, 2.5 mg, 10 mg etc) and ii) the first week and the remaining weeks for each study period
Time spent above various thresholds of beta-hydroxybutyrate concentrations: | 17 weeks
  ≥ 0.3 mmol/L, ≥ 0.6 mmol/L, ≥ 0.8 mmol/L ≥ 1.5 mmol/L, ≥ 3.0 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tsoukas, M.D., Principal Investigator — Clinique Medicale Hygea
Locations (1):
- Hygea Medical Clinic, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data and informed consent form will be shared by the corresponding author, for academic purposes, subject to a material transfer agreement and approval of the McGill University Health Center's Research Ethics Board. All data shared will be de-identified. Raw data will be shared for non-commercial use upon reasonable request and a material transfer agreement.
Supporting Information: ICF